CLINICAL TRIAL: NCT06304870
Title: Impact of Blocking the Glossopharyngeal Nerve on Gastroesophageal Reflux Disease: A Randomized Double-blind Controlled Study
Brief Title: Impact of Blocking the Glossopharyngeal Nerve on Gastroesophageal Reflux Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad (Other)
Responsible Party: Sponsor-Investigator, Muhammad, Research Director, Ahmadu Bello University Teaching Hospital
Organization: Ahmadu Bello University Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYB-reflux
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Rehabilitation; Lidocaine; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation therapy+Placebo Glossopharyngeal Nerve Block (Placebo Comparator): The study lasts 20d for each patient. During the treatment, All the participants are provided with the rehabilitation therapy and placebo nerve block.
  Interventions: Behavioral: Rehabilitation therapy; Procedure: Injection
- Rehabilitation therapy+Glossopharyngeal Nerve Block (Experimental): The study lasts 20d for each patient. During the treatment, All the participants are provided with the rehabilitation therapy. Based on this, the patients in the experimental group are provided with Stellate Ganglion Block , using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g), once a day.
  Interventions: Behavioral: Rehabilitation therapy; Drug: Lidocaine; Procedure: Injection

INTERVENTIONS:
Behavioral: Rehabilitation therapy — Rehabilitation therapy includes Diet management: Avoiding consumption of irritant foods and beverages, such as spicy foods, caffeine, alcohol, and acidic foods. Controlling portion sizes and meal timing, and adopting smaller, more frequent meals.
  Lifestyle adjustments: Avoiding lying down or bending immediately after meals, maintaining a sitting or upright position for at least 2 hours. Adjusting sleeping positions by elevating the head of the bed to reduce nighttime acid reflux. Avoiding excessive exertion and managing stress levels.
  Rehabilitation training: Strengthening the control of esophageal and gastric muscles through rehabilitation exercises to improve the function of the gastroesophageal sphincter and prevent gastric fluid reflux.
Drug: Lidocaine — The patient lies supine without a pillow, turns the head to the contralateral side of the block, and at the midpoint of the line connecting the angle of the mandible with the mastoid process (the styloid process), the skin is disinfected, and a 22-gauge, 3.8 cm puncture needle is loaded onto a 5 mL syringe. The puncture needle is inserted perpendicularly to the skin surface at the styloid process, and advanced through the skin and subcutaneous tissue until it contacts the bone of the styloid process. The puncture needle is then retracted and advanced anteriorly beyond the styloid process by 0.5-1.0 cm. When no blood or cerebrospinal fluid is aspirated, the blocking drug can be injected [20 g/L lidocaine injection].
  Arms: Rehabilitation therapy+Glossopharyngeal Nerve Block
Procedure: Injection — The patient lies supine without a pillow, turns the head to the contralateral side of the block, and at the midpoint of the line connecting the angle of the mandible with the mastoid process (the styloid process), the skin is disinfected, and a 22-gauge, 3.8 cm puncture needle is loaded onto a 5 mL syringe. The puncture needle is inserted perpendicularly to the skin surface at the styloid process, and advanced through the skin and subcutaneous tissue until it contacts the bone of the styloid process.

SUMMARY:
The goal of this clinical trial is to explore Clinical Effect of Glossopharyngeal Nerve Block on Pharyngeal Dysphagia Induced by Gastroesophageal Reflux Disease. The main question it aims to answer is:

• Can Glossopharyngeal Nerve Block improve dysphagia caused by gastroesophageal reflux symptoms on the basis of rehabilitation training? Participants will be randomly allocated into the control group or the experimental group, all under rehabilitation treatment, the experimental group will be given Glossopharyngeal Nerve Block once a day additionally. The study lasts 20 days for each participant. Researchers will compare the Rosenbek penetration-aspiration scale, Gastroesophageal Reflux Disease Questionnaire, Pressure pain threshold, to see if the Glossopharyngeal Nerve Block can help improve the symptom.

DETAILED DESCRIPTION:
Gastroesophageal reflux is a common digestive disorder characterized by the backflow of stomach contents and fluids into the esophagus.

The goal of this clinical trial is to explore Clinical Effect of Glossopharyngeal Nerve Block on Pharyngeal Dysphagia Induced by Gastroesophageal Reflux Disease. The main question it aims to answer is:

• Can Glossopharyngeal Nerve Block improve dysphagia caused by gastroesophageal reflux symptoms on the basis of rehabilitation training? Participants will be randomly allocated into the control group or the experimental group, all under rehabilitation treatment, the experimental group will be given Glossopharyngeal Nerve Block once a day additionally. The study lasts 20 days for each participant. Researchers will compare the Rosenbek penetration-aspiration scale, Gastroesophageal Reflux Disease Questionnaire, Pressure pain threshold, to see if the Glossopharyngeal Nerve Block can help improve the symptom.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic criteria for Gastroesophageal Reflux Disease.
* Age between 18 and 65 years.
* Confirmed tongue-pharyngeal nerve injury by electromyography.
* Esophageal manometry and barium swallow examination confirming the presence of pharyngeal dysphagia.
* Normal higher brain function, able to cooperate with treatment.

Exclusion Criteria:

* Brain vascular disease diagnosed.
* Clinical assessment and swallowing videofluoroscopic examination revealing cognitive phase, oral preparatory phase, or oral phase disorders.
* Concurrent presence of other neurological disorders such as Alzheimer's disease, traumatic brain injury, Parkinson's disease.
* Esophageal obstruction and severe liver or kidney dysfunction
* Subjective unwillingness to undergo the treatment and presence of psychiatric abnormalities, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Rosenbek penetration-aspiration scale | day 1 and day 20
  This assessment evaluated the patient's swallowing of contrast medium and whether there was retention, penetration, and aspiration. It included multiple items, each with the corresponding criteria, Specifically, whether the swallowed material entered the airway, passed through or contacted the vocal cords, and whether the patient exhibited the corresponding ability to clear. There were 8 levels in the results, with higher levels indicating more severe aspiration.

SECONDARY OUTCOMES:
Gastroesophageal Reflux Disease Questionnaire | day 1 and day 20
  The Gastroesophageal Reflux Disease Questionnaire is a commonly used questionnaire for assessing the symptoms and severity of gastroesophageal reflux disease. It was developed by gastrointestinal experts in Germany and consists of six questions that evaluate the frequency and severity of gastroesophageal reflux disease symptoms. The maximum score for the Test is 12 points, with a lower score indicating milder symptoms and a higher score indicating more severe symptoms.
Pressure pain threshold | day 1 and day 20
  Pressure is applied on the spinous processes of the fourth cervical vertebrae. Pressure will be uniformly increased, and patients are given the identical instruction, "let me know when the sensation of pressure becomes uncomfortable or painful". At this point, the pressure will be immediately released, and the plunger is retracted by the evaluator. And the pressure will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Principal Investigator — Site Coordinator of United Medical Group

IPD SHARING:
Plan to Share IPD: No